CLINICAL TRIAL: NCT05783076
Title: Stereotactic Body Radiation Therapy and vNKT Cell Adoptive Therapy for Advanced Pancreatic Cancer: a Phase 2 Trial
Brief Title: SBRT Plus vNKT for Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhang Huo Jun, Professor, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChangHai PDAC
Record Dates: First submitted 2023-03-02; First posted 2023-03-24 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery; Radiotherapy; Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stereotactic body radiation therapy plus vNKT cells (Experimental): Stereotactic body radiatuon therapy is performed by Cyberknife, an image-guided frameless stereotactic robotic radiosurgery system (Accuray Corporation, Sunnyvale CA). Prescription doses ranged from 35-40Gy/5f.
  Allogeneic peripherial blood monocytes (PBMC) are collected from healthy individuals. vNKT cells are isolated from PBMC and then expanded. Quality tests shoud be performed before isolated cells become cell therapy products. After quality control, vNKT cells should be transfused into patients within 24 hours. Adoptive cell therapy is initiated 2-3 weeks after SBRT. Cell therapy is performed twice a month with the interval of 24-48 hours within 6 months after SBRT. The number of vNKT cells transfused once is 1.5×10^8/Kg±15%. While cell therapy is performed once a months 6 months after SBRT. Cell therapy will be delivered for one year or until disease progression if it occurs within one year.
  Interventions: Drug: Stereotactic body radiation therapy; Drug: adoptive cell therapy with vNKT cells

INTERVENTIONS:
Drug: Stereotactic body radiation therapy — Details have been shown in arm descriptions.
  Other Names: Radiotherapy
Drug: adoptive cell therapy with vNKT cells — Details have been shown in arm descriptions.
  Other Names: adoptive cell therapy

SUMMARY:
Owing to that the previous study of the investigators showed that SBRT plus pembrolizumab and trametinib provided favorable outcomes compared with SBRT plus gemcitabine for pancreatic cancer, therefore, the investigators aim to further investigate the efficacy and safety of SBRT plus another kind of immunotherapy, namely adoptive cell therapy (vNKT cell), for advanced pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer still remains one of the most lethal malignancies and fourth leading cancer cause of death in US, with a slight increasing incidence and the lowest 5-year survival rate of 9%. Although surgical resection is considered as the radical treatment, most patients were not amenable to surgery due to the initial diagnosis of advanced pancreatic cancer. For those patients, stereotactic body radiation therapy (SBRT), recommended as the local treatment, combining with chemotherapy is the optimal treatment. Despite improved knowledge about the genetic background and an increasing understanding of the tumor microenvironment, immunotherapy especially immune checkpoint inhibitors, although efficient for many solid malignancies, including metastatic melanoma and lung cancer, have not yielded any clinical benefit in pancreatic cancer.

In addition to immune checkpoint inhibitors, chimeric antigen receptor T cell (CAR-T) has shown promising efficacy in hematologic malignancies. Nowadays, adoptive cell therapy includes CD8+ T cells and NK cells modified with chimeric antigen receptors. However, due to limited technology, expansion of specific CD8+ T cells is quite difficult. Additionally, there is lack of specific tumor antigens in solid tumors, which results in unsatisfactory outcomes of CAR-T and CAR-NK cells targeting solid tumors. Therefore, novel cell therapies may provide insights into therapies for solid tumors. Recently, vNKT and γδT cells used in trials of cell therapy have aroused attention.

NKT cells possess both phenotypes of T cells and NK cells. Hence, NKT cells could secret various cytokines and chemokines after stimulations to enhance anti-tumor immunity independent of MHC. Also, cytotoxic effects of NKT cells could be activated via T cell receptors (TCR) targeting specific antigens. There are two kinds of NKT cells. One is classic NKT cells with invariant TCR which are specialized CD1d-restricted T cells that recognize lipid antigens, called iNKT (invariant NKT) cells. The other is non-CD1d-restrcited. This CD8+ NKT cells has more potent anti-tumor effects than conventional T and NK cells, which is manifested by killing tumor cells and myeloid derived suppressor cells. Owing to recognition of MHC-restricted antigens via diverse TCRs, they are called vNKT (variant NKT) cells.

Furthermore, our previous studies has clarified favorable outcomes from the synergy of SBRT plus immunotherapy for pancreatic cancer. Therefore, the investigators aim to investigate the efficacy and safety of SBRT plus vNKT cell adoptive therapy for advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years.
2. Pathological confirmed pancreatic ductal adenocarcinoma.
3. No previous immunotherapy or radiotherapy, or more than one year after the last course of radiotherapy.
4. History of sugery or chemotherapy, and documented disease progressions after these therapies.
5. ECOG performance status of 0-2 points.
6. Normal results of laboratory tests, including WBC ≥4.0×10^9/L, Neu ≥2.0×10^9/L, Hb ≥120g/L, Plt ≥100×10^9/L; AST, ALT <2.5 times of the upper limit of normal, total bilirubin <17.1μmol/L, creatinine <110μmoI/L; international normalized ratio in coagulation test <2.0
7. Willing to participate in the study and complete follow-up examinations as required.

Exclusion Criteria:

1. History of immunotherapy, or less than one year after the last course of radiotherapy.
2. History of other tumors.
3. Confirmed synchronous multiple tumors.
4. ECOG performance status of more than 2 points.
5. Active inflammatory bowel disease, or peptic ulcer.
6. History of gastrointestinal bleeding or perforation within 6 months.
7. Infections required antibiotics.
8. Positive HBsAg or HCV antibody.
9. Positive HIV antibody.
10. Impaired heart function (NYHA III-IV level), respiratory insufficiency.
11. Confirmed genetic diseases.
12. History of hematologic diseases, including leukemia, lymphoma, myeloma or myelodysplastic syndrome.
13. History of stem cell or organ transplantation.
14. History of autoimmune diseases except leukoderma punctata.
15. Severe anaphylaxis.
16. Long term use of immunosuppressors or steroids.
17. Receiving chemotherapy at the time of screening stage, or participation of other studies.
18. Pregnancy or lactation.
19. Unable to understand the whole procedure of study and provide written informed consent.
20. No comprehensive understanding about patients' immune functions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-06-25 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival will be determined | From randomization to death irrespective of cause, assessed up to 2 years
  From randomization to death irrespective of cause

SECONDARY OUTCOMES:
Progression free survival will be determined | From randomization to documentation of any clinical or radiological disease progression or death, whichever occurred first, assessed up to 2 years
  From randomization to documentation of any clinical or radiological disease progression or death, whichever occurred first
Adverse effects will be determined | Up to 2 years
  Assessed according to the National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE; version 4.0)
Quality of life will be determined | Up to 2 years
  Assessed with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30. The score of each scale ranges from 0 to 100. Higher scores in function domains and global health status indicate better quality of life, while higher scores in symptom domains imply worse quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital affiliated to Naval Medical University, Shanghai, China

REFERENCES:
- [Derived] Zhu X, Yin X, Liu W, Yu C, Xia S, Cao Y, Jiang L, Guo Z, Zhang M, Zhang H. Stereotactic body radiation therapy plus adoptive vNKT cell therapy for pancreatic cancer: protocol of a phase II trial. Immunotherapy. 2025 Jul;17(10):685-692. doi: 10.1080/1750743X.2025.2533112. Epub 2025 Jul 16. PMID 40671381